CLINICAL TRIAL: NCT01263314
Title: A Single Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of MK-8266 in Elderly Subjects With Hypertension
Brief Title: Safety, Tolerability, and Pharmacokinetics of MK-8266 in Elderly Participants With High Blood Pressure (MK-8266-003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8266-003; MK-8266-003 (Other: Merck Protocol Number)
Record Dates: First submitted 2010-11-15; First posted 2010-12-20 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-03

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Panel A MK-8266 0.3 mg (Elderly Males with Mild/Mod. HTN) (Experimental): MK-8266 single dose 0.3 mg
  Interventions: Drug: MK-8266
- Panel A MK-8266 0.6 mg (Elderly Males with Mild/Mod. HTN) (Experimental): MK-8266 single dose 0.6 mg
  Interventions: Drug: MK-8266
- Panel A MK-8266 0.7/0.3 mg (Elderly Males with Mild/Mod. HTN) (Experimental): MK-8266 single dose 0.7 mg and then 0.3 mg after 10 hours
  Interventions: Drug: MK-8266
- Panel A Placebo to MK-8266 (Elderly Males with Mild/Mod. HTN) (Placebo Comparator): Placebo to MK-8266 single dose
  Interventions: Drug: Placebo
- Panel B MK-8266 0.3 mg (Elderly Females with Mild/Mod. HTN) (Experimental): MK-8266 single dose 0.3 mg
  Interventions: Drug: MK-8266
- Panel B MK-8266 0.6 mg (Elderly Females with Mild/Mod. HTN) (Experimental): MK-8266 single dose 0.6 mg
  Interventions: Drug: MK-8266
- Panel B MK-8266 0.7/0.3 mg (Elderly Fem. with Mild/Mod. HTN) (Experimental): MK-8266 single dose 0.7 mg and then 0.3 mg after 10 hours
  Interventions: Drug: MK-8266
- Panel B Placebo to MK-8266 (Elderly Fem. with Mild/Mod. HTN) (Placebo Comparator): Placebo to MK-8266 single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-8266 — Oral capsules, 0.1 mg potency
  Arms: Panel A MK-8266 0.3 mg (Elderly Males with Mild/Mod. HTN); Panel A MK-8266 0.6 mg (Elderly Males with Mild/Mod. HTN); Panel A MK-8266 0.7/0.3 mg (Elderly Males with Mild/Mod. HTN); Panel B MK-8266 0.3 mg (Elderly Females with Mild/Mod. HTN); Panel B MK-8266 0.6 mg (Elderly Females with Mild/Mod. HTN); Panel B MK-8266 0.7/0.3 mg (Elderly Fem. with Mild/Mod. HTN)
Drug: Placebo — Oral placebo capsules to match MK-8266 capsules
  Arms: Panel A Placebo to MK-8266 (Elderly Males with Mild/Mod. HTN); Panel B Placebo to MK-8266 (Elderly Fem. with Mild/Mod. HTN)

SUMMARY:
This is a randomized, double-blind, placebo-controlled study. The hypothesis for this study is that single oral doses of MK-8266 selected for this study are sufficiently safe and well tolerated by elderly male and elderly female participants with hypertension to permit continued clinical investigation.

DETAILED DESCRIPTION:
Two panels, each consisting of eight participants (8 elderly males with mild to moderate hypertension in Panel A and 8 elderly females with mild to moderate hypertension in Panel B) will be randomized to receive either MK-8266 or matching placebo in a 3:1 ratio. Participants will receive single doses of MK-8266 or matching placebo in three treatment periods (Periods 1 through 3). In both Panel A and Panel B, doses will escalate in a rising, fixed sequence. In Period 1 (0.3 mg), Period 2 (0.6 mg), and Period 3 (0.7 mg and then 0.3 mg 10 hours later) once daily doses of MK-8266 or matching placebo will be administered.

All participants will receive at least 2 doses of MK-8266. Participants completing placebo treatment in Period 1 will flow to the MK-8266 arm in the next period, with 2 participants from the MK-8266 arm receiving placebo in the next period.

Blood samples will be obtained pre-dose and at selected time points up to 48 hours post-dose for determination of MK-8266 plasma concentrations.

ELIGIBILITY:
Inclusion criteria:

* Participants are male or non-childbearing female.
* Participant with essential hypertension (HTN), Grade 1 or 2 (as per European Society of Hypertension [ESH]) or isolated mild to moderate systolic HTN. High normal systolic BP ≥130 mmHg will be also allowed. Blood pressures to be confirmed on at least three occasions pre-study. The possibility of secondary causes of HTN should be assessed. Participants who are being treated for HTN with drugs (including beta blocking medications) may be able to participate if the drug doses can be reduced or discontinued, at the discretion of the investigator.
* Participants with a Body Mass Index (BMI) ≤35 kg/m^2 at the screening visit.
* Participants judged to be generally in good health based on medical history, physical examination, vital sign measurements (with the exception of HTN), and laboratory safety tests performed at the screening visit.
* Participant has no clinically significant abnormality (confirmed by the investigator in consultation with the Merck Clinical Monitor) on electrocardiogram (ECG) or Holter Monitor Evaluation performed at the screening visit and/or prior to administration of the initial dose of study drug.
* Participants must have a platelet count ≥150,000 cu/mL at the screening and pre-study visit.
* Participants, at screening, will have a positive Augmentation Index.
* Participant has been a nonsmoker and/or has not used nicotine or nicotine-containing products for at least 6 months; participants who have discontinued smoking or the use of nicotine/nicotine containing products for at least 3 months may be enrolled at the discretion of the investigator.
* Participant is willing to comply with the study restrictions.
* Participant has a negative test for hidden blood in the stool at screening.

Exclusion criteria:

* Participants who have had situational depression may be enrolled in the study at the discretion of the investigator.
* Participant has an estimated creatinine clearance of ≤60 mL/min based on the Cockcroft-Gault equation.
* Participant has a history of stroke, chronic seizures, or major neurological disorder.
* Participant has a history of clinically significant endocrine, gastrointestinal, cardiovascular (with the exception of HTN), hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases. Participants with a history of uncomplicated kidney stones or childhood asthma may be enrolled in the study at the discretion of the investigator.
* Patient demonstrates low blood pressure at screening and Pre-dose Day 1 while going from a semi-recumbent to standing position.
* Participant has a functional disability that can interfere with rising from a semi-recumbent position to the standing position.
* Participant has any personal or family history of a bleeding or a clotting disorder.
* Participant has a history of frequent nosebleeds.
* Participant has a history of cancer with the exceptions of: adequately treated non-melanoma skin carcinoma or carcinoma in situ of the cervix; other malignancies which have been successfully treated >10 years prior to the screening visit, for which in the judgment of both the investigator and treating physician, appropriate follow-up has revealed no evidence of recurrence from the time of treatment through the time of the screening visit; or, participants, who, in the opinion of the study investigator, are highly unlikely to sustain a recurrence for the duration of the study.
* Participant has a history of clinically significant cardiac disease including, but not limited to hemodynamically relevant heart valve disease (if there would be any uncertainty about the diagnosis, confirmation with an echocardiography within 3 months of screening is required), or evidence of secondary cardiac damage.
* Participant is categorized as a class II or greater functional classification for heart failure according to the New York Heart Association (NYHA).
* Participant is unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs or herbal remedies (such as St. John's Wort [Hypericum perforatum]) beginning approximately 2 weeks (or 5 half-lives) prior to administration of the initial dose of study drug, throughout the study until the post-study visit. Certain medication use may be permitted after consultation with the Merck clinical monitor.
* Participant currently and regularly uses aspirin (including low dose) and cannot be discontinued from it from 2 weeks prior to study start or has used aspirin within 2 weeks prior to study start (and anticipates using it during the course of the study); this applies also to any pain relievers and cold or sinus remedies that have aspirin in them, and the use of anti-platelet drugs, such as clopidogrel or dipyridamole. Chronic use of certain non-steroidal anti-inflammatory drugs (NSAIDs) such as ≥500 mg of naproxen twice a day must be also avoided beginning at least 2 weeks prior the study and until the post-study visit.
* Participant anticipates using sildenafil (Viagra®), tadalafil (Cialis®), or Vardenafil (Levitra®).
* Participant uses or anticipates using organic nitrate preparations (for example, nitroglycerin, isosorbide mononitrate, isosorbide dinitrate or pentaerythritol) during the course of the study.
* Participant consumes excessive amounts of alcohol, defined as greater than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [284 mL/10 ounces], wine [125 mL/4 ounces], or distilled spirits [25 mL/1 ounce]) per day. Participants that consume 4 glasses of alcoholic beverages per day may be enrolled at the discretion of the investigator.
* Participant consumes excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, or other caffeinated beverages per day.
* Participant has had major surgery, donated or lost 1 unit of blood (approximately 500 mL) or participated in another investigational study within 4 weeks prior to the screening visit. The 4-week window will be derived from the date of the last study procedure (i.e., post-study, AE follow-up, etc.) in the previous study to the screening visit of the current study.
* Participant has a history of significant multiple and/or severe allergies (including latex allergy), or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food.
* Participant is currently a regular user of illicit drugs or has a history of drug/alcohol abuse within approximately 1 year of the screening visit.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-11-01 (Actual); Primary Completion 2011-02-01 (Actual); Study Completion 2011-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants will receive at least 2 doses of MK-8266. Participants completing placebo treatment in Period 1 will flow to the MK-8266 arm in the next period, with 2 participants from the MK-8266 arm receiving placebo in the next period.
Groups:
- Panel A (Elderly Males, Mild/Moderate Hypertension) Sequence 1; Panel B (Elderly Females, Mild/Moderate Hypertension) Seq. 2: Period 1: MK-8266 0.3 mg; Period 2: MK-8266 0.6 mg; and Period 3: placebo.
- Panel A (Elderly Males, Mild/Moderate Hypertension) Sequence 2; Panel B (Elderly Females, Mild/Moderate Hypertension) Seq. 3: Period 1: MK-8266 0.3 mg; Period 2: MK-8266 0.6 mg; and Period 3: MK-8266 0.7 mg and then 0.3 mg after 10 hours.
- Panel A (Elderly Males, Mild/Moderate Hypertension) Sequence 3; Panel B (Elderly Females, Mild/Moderate Hypertension) Seq. 1: Period 1: MK-8266 0.3 mg; Period 2: placebo; and Period 3: MK-8266 0.7 mg and then 0.3 mg after 10 hours.
- Panel A (Elderly Males, Mild/Moderate Hypertension) Sequence 4; Panel B (Elderly Females, Mild/Moderate Hypertension) Seq. 4: Period 1: placebo; Period 2: MK-8266 0.6 mg; and Period 3: MK-8266 0.7 mg and then 0.3 mg after 10 hours.
Period: Period 1
Arm/Group | Panel A (Elderly Males, Mild/Moderate Hypertension) Sequence 1 | Panel A (Elderly Males, Mild/Moderate Hypertension) Sequence 2 | Panel A (Elderly Males, Mild/Moderate Hypertension) Sequence 3 | Panel A (Elderly Males, Mild/Moderate Hypertension) Sequence 4 | Panel B (Elderly Females, Mild/Moderate Hypertension) Seq. 1 | Panel B (Elderly Females, Mild/Moderate Hypertension) Seq. 2 | Panel B (Elderly Females, Mild/Moderate Hypertension) Seq. 3 | Panel B (Elderly Females, Mild/Moderate Hypertension) Seq. 4
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Panel A (Elderly Males, Mild/Moderate Hypertension) Sequence 1 | Panel A (Elderly Males, Mild/Moderate Hypertension) Sequence 2 | Panel A (Elderly Males, Mild/Moderate Hypertension) Sequence 3 | Panel A (Elderly Males, Mild/Moderate Hypertension) Sequence 4 | Panel B (Elderly Females, Mild/Moderate Hypertension) Seq. 1 | Panel B (Elderly Females, Mild/Moderate Hypertension) Seq. 2 | Panel B (Elderly Females, Mild/Moderate Hypertension) Seq. 3 | Panel B (Elderly Females, Mild/Moderate Hypertension) Seq. 4
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Panel A (Elderly Males, Mild/Moderate Hypertension) Sequence 1 | Panel A (Elderly Males, Mild/Moderate Hypertension) Sequence 2 | Panel A (Elderly Males, Mild/Moderate Hypertension) Sequence 3 | Panel A (Elderly Males, Mild/Moderate Hypertension) Sequence 4 | Panel B (Elderly Females, Mild/Moderate Hypertension) Seq. 1 | Panel B (Elderly Females, Mild/Moderate Hypertension) Seq. 2 | Panel B (Elderly Females, Mild/Moderate Hypertension) Seq. 3 | Panel B (Elderly Females, Mild/Moderate Hypertension) Seq. 4
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics for all participants receiving study treatment. Participants are grouped according to either Panel A or Panel B (i.e. males or females with mild/moderate hypertension).
Groups:
- Panel A (Elderly Males, Mild/Moderate Hypertension); Panel B (Elderly Females, Mild/Moderate Hypertension): MK-8266 (0.3 mg, 0.6 mg, or 0.7 mg and then 0.3 mg after 10 hours) or placebo
- Total: Total of all reporting groups
Arm/Group | Panel A (Elderly Males, Mild/Moderate Hypertension) | Panel B (Elderly Females, Mild/Moderate Hypertension) | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.0 (2.8) | 68.9 (2.8) | 68.4 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 8 | 8
  Male | 8 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to 48 days
Population: All participants who received at least one dose of the investigational drug.
Measure: Count of Participants; unit: Participants
Groups:
- Panel A MK-8266 0.3 mg (Elderly Males With Mild/Moderate HTN): MK-8266 single dose 0.3 mg
  Hypertension (HTN)
- Panel A MK-8266 0.6 mg (Elderly Males With Mild/Moderate HTN); Panel B MK-8266 0.6 mg (Elderly Females, Mild/Moderate HTN): MK-8266 single dose 0.6 mg
- Panel A MK-8266 0.7 /0.3 mg (Elderly Males, Mild/Moderate HTN); Panel B MK-8266 0.7/0.3 mg (Elderly Fem., Mild/Moderate HTN): MK-8266 0.7 mg and then 0.3 mg after 10 hours
- Panel A Placebo to MK-8266 (Elderly Males, Mild/Moderate HTN); Panel B Placebo to MK-8266 (Elderly Fem., Mild/Moderate HTN): Placebo to MK-8266 single dose
- Panel B MK-8266 0.3 mg (Elderly Females, Mild/Moderate HTN): MK-8266 single dose 0.3 mg
Arm/Group | Panel A MK-8266 0.3 mg (Elderly Males With Mild/Moderate HTN) | Panel A MK-8266 0.6 mg (Elderly Males With Mild/Moderate HTN) | Panel A MK-8266 0.7 /0.3 mg (Elderly Males, Mild/Moderate HTN) | Panel A Placebo to MK-8266 (Elderly Males, Mild/Moderate HTN) | Panel B MK-8266 0.3 mg (Elderly Females, Mild/Moderate HTN) | Panel B MK-8266 0.6 mg (Elderly Females, Mild/Moderate HTN) | Panel B MK-8266 0.7/0.3 mg (Elderly Fem., Mild/Moderate HTN) | Panel B Placebo to MK-8266 (Elderly Fem., Mild/Moderate HTN)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 4 | 4 | 3 | 1 | 5 | 4 | 4 | 4

2. Primary Outcome: Number of Participants With Abnormal Laboratory Hematology Values Reported as an AE
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. Abnormal laboratory hematology value was any AE reported under the System Organ Class of Investigations that was related to an abnormal laboratory hematology value.
Time Frame: Up to 48 days
Population: All participants who received at least one dose of the investigational drug.
Measure: Count of Participants; unit: Participants
Groups:
- Panel A MK-8266 0.3 mg (Elderly Males With Mild/Moderate HTN); Panel B MK-8266 0.3 mg (Elderly Females, Mild/Moderate HTN): MK-8266 single dose 0.3 mg
Arm/Group | Panel A MK-8266 0.3 mg (Elderly Males With Mild/Moderate HTN) | Panel A MK-8266 0.6 mg (Elderly Males With Mild/Moderate HTN) | Panel A MK-8266 0.7 /0.3 mg (Elderly Males, Mild/Moderate HTN) | Panel A Placebo to MK-8266 (Elderly Males, Mild/Moderate HTN) | Panel B MK-8266 0.3 mg (Elderly Females, Mild/Moderate HTN) | Panel B MK-8266 0.6 mg (Elderly Females, Mild/Moderate HTN) | Panel B MK-8266 0.7/0.3 mg (Elderly Fem., Mild/Moderate HTN) | Panel B Placebo to MK-8266 (Elderly Fem., Mild/Moderate HTN)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Abnormal Laboratory Chemistry Values Reported as an AE
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. Abnormal laboratory chemistry value was any AE reported under the System Organ Class of Investigations that was related to an abnormal laboratory chemistry value.
Time Frame: Up to 48 days
Population: All participants who received at least one dose of the investigational drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Panel A MK-8266 0.3 mg (Elderly Males With Mild/Moderate HTN) | Panel A MK-8266 0.6 mg (Elderly Males With Mild/Moderate HTN) | Panel A MK-8266 0.7 /0.3 mg (Elderly Males, Mild/Moderate HTN) | Panel A Placebo to MK-8266 (Elderly Males, Mild/Moderate HTN) | Panel B MK-8266 0.3 mg (Elderly Females, Mild/Moderate HTN) | Panel B MK-8266 0.6 mg (Elderly Females, Mild/Moderate HTN) | Panel B MK-8266 0.7/0.3 mg (Elderly Fem., Mild/Moderate HTN) | Panel B Placebo to MK-8266 (Elderly Fem., Mild/Moderate HTN)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Abnormal Laboratory Urinalysis Values Reported as an AE
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. Abnormal laboratory urinalysis value was any AE reported under the System Organ Class of Investigations that was related to an abnormal laboratory urinalysis value.
Time Frame: Up to 37 days
Population: All participants who received at least one dose of the investigational drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Panel A MK-8266 0.3 mg (Elderly Males With Mild/Moderate HTN) | Panel A MK-8266 0.6 mg (Elderly Males With Mild/Moderate HTN) | Panel A MK-8266 0.7 /0.3 mg (Elderly Males, Mild/Moderate HTN) | Panel A Placebo to MK-8266 (Elderly Males, Mild/Moderate HTN) | Panel B MK-8266 0.3 mg (Elderly Females, Mild/Moderate HTN) | Panel B MK-8266 0.6 mg (Elderly Females, Mild/Moderate HTN) | Panel B MK-8266 0.7/0.3 mg (Elderly Fem., Mild/Moderate HTN) | Panel B Placebo to MK-8266 (Elderly Fem., Mild/Moderate HTN)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP)
Description: Participants rested for at least 10 minutes prior to having vital sign measurements obtained.
Time Frame: Baseline and 0 to 8 hours postdose
Population: All participants who received at least one dose of the investigational drug.
Measure: Least Squares Mean (Standard Deviation); unit: Millimeters of mercury
Groups:
- Panel A MK-8266 0.7 /0.3 (Elderly Males With Mild/Mod. HTN); Panel B MK-8266 0.7/0.3 mg (Elderly Fem., Mild/Moderate HTN): MK-8266 0.7 mg and then 0.3 mg after 10 hours
- Panel A Placebo to MK-8266 (Elderly Males Mild/Moderate HTN): Placebo to MK- 8266 single dose
Arm/Group | Panel A MK-8266 0.3 mg (Elderly Males With Mild/Mod. HTN) | Panel A MK-8266 0.6 mg (Elderly Males With Mild/Mod. HTN) | Panel A MK-8266 0.7 /0.3 (Elderly Males With Mild/Mod. HTN) | Panel A Placebo to MK-8266 (Elderly Males Mild/Moderate HTN) | Panel B MK-8266 0.3 mg (Elderly Females With Mild/Mod. HTN) | Panel B MK-8266 0.6 mg (Elderly Females, Mild/Moderate HTN) | Panel B MK-8266 0.7/0.3 mg (Elderly Fem., Mild/Moderate HTN) | Panel B Placebo to MK-8266 (Elderly Fem., Mild/Moderate HTN)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Millimeters of mercury
  Baseline | 148.3 (8.87) | 137.2 (19.09) | 134.0 (12.96) | 132.7 (10.93) | 141.7 (13.38) | 139.5 (11.10) | 137.7 (7.76) | 142.0 (18.10)
  Change from Baseline | -0.71 (3.85) | -0.79 (7.44) | -1.13 (4.13) | 0.54 (4.83) | -0.33 (10.01) | -4.16 (10.25) | -2.28 (5.87) | 5.91 (9.00)
Statistical Analysis 1: Comparison: Panel A MK-8266 0.3 mg (Elderly Males With Mild/Mod. HTN) vs Panel A Placebo to MK-8266 (Elderly Males Mild/Moderate HTN); Test type: Other; p = 0.3551, ANOVA; Mean Difference (Final Values) = -1.25, 90% CI 2-sided [-7.01 to 4.50]
Statistical Analysis 2: Comparison: Panel A MK-8266 0.6 mg (Elderly Males With Mild/Mod. HTN) vs Panel A Placebo to MK-8266 (Elderly Males Mild/Moderate HTN); Test type: Other; p = 0.3474, ANOVA; Mean Difference (Final Values) = -1.32, 90% CI 2-sided [-7.08 to 4.48]
Statistical Analysis 3: Comparison: Panel A MK-8266 0.7 /0.3 (Elderly Males With Mild/Mod. HTN) vs Panel A Placebo to MK-8266 (Elderly Males Mild/Moderate HTN); Test type: Other; p = 0.3105, ANOVA; Mean Difference (Final Values) = -1.67, 90% CI 2-sided [-7.42 to 4.09]
Statistical Analysis 4: Comparison: Panel B MK-8266 0.3 mg (Elderly Females With Mild/Mod. HTN) vs Panel B Placebo to MK-8266 (Elderly Fem., Mild/Moderate HTN); Test type: Other; p = 0.1346, ANOVA; Mean Difference (Final Values) = -6.25, 90% CI 2-sided [-15.8 to 3.27]
Statistical Analysis 5: Comparison: Panel B MK-8266 0.6 mg (Elderly Females, Mild/Moderate HTN) vs Panel B Placebo to MK-8266 (Elderly Fem., Mild/Moderate HTN); Test type: Other; p = 0.0416, ANOVA; Mean Difference (Final Values) = -10.1, 90% CI 2-sided [-19.6 to -0.56]
Statistical Analysis 6: Comparison: Panel B MK-8266 0.7/0.3 mg (Elderly Fem., Mild/Moderate HTN) vs Panel B Placebo to MK-8266 (Elderly Fem., Mild/Moderate HTN); Test type: Other; p = 0.0762, ANOVA; Mean Difference (Final Values) = -8.20, 90% CI 2-sided [-17.7 to 1.32]

6. Primary Outcome: Change From Baseline in Heart Rate
Description: Participants rested for at least 10 minutes prior to having vital sign measurements obtained. Heart rate measurements were obtained in the semirecumbent position and 3 sets of measurements were obtained approximately 1 minute apart.
Time Frame: Baseline and 0 to 8 hours postdose
Population: All participants who received at least one dose of the investigational drug.
Measure: Least Squares Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Panel A MK-8266 0.3 mg (Elderly Males With Mild/Mod. HTN) | Panel A MK-8266 0.6 mg (Elderly Males With Mild/Mod. HTN) | Panel A MK-8266 0.7 /0.3 (Elderly Males With Mild/Mod. HTN) | Panel A Placebo to MK-8266 (Elderly Males Mild/Moderate HTN) | Panel B MK-8266 0.3 mg (Elderly Females With Mild/Mod. HTN) | Panel B MK-8266 0.6 mg (Elderly Females, Mild/Moderate HTN) | Panel B MK-8266 0.7/0.3 mg (Elderly Fem., Mild/Moderate HTN) | Panel B Placebo to MK-8266 (Elderly Fem., Mild/Moderate HTN)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Beats per minute
  Baseline | 68.83 (9.24) | 67.83 (10.53) | 58.33 (5.50) | 69.00 (8.37) | 65.33 (5.32) | 65.00 (5.97) | 61.33 (4.23) | 63.83 (5.64)
  Change from Baseline | 0.58 (6.12) | 4.23 (4.78) | 7.90 (4.89) | 0.11 (7.85) | 2.40 (2.37) | 5.51 (3.27) | 6.65 (3.33) | 1.25 (3.57)
Statistical Analysis 1: Comparison: Panel A MK-8266 0.3 mg (Elderly Males With Mild/Mod. HTN) vs Panel A Placebo to MK-8266 (Elderly Males Mild/Moderate HTN); Test type: Other; p = 0.418, ANOVA; Mean Difference (Final Values) = 0.47, 90% CI 2-sided [-3.47 to 4.41]
Statistical Analysis 2: Comparison: Panel A MK-8266 0.6 mg (Elderly Males With Mild/Mod. HTN) vs Panel A Placebo to MK-8266 (Elderly Males Mild/Moderate HTN); Test type: Other; p = 0.0434, ANOVA; Mean Difference (Final Values) = 4.12, 90% CI 2-sided [0.18 to 8.05]
Statistical Analysis 3: Comparison: Panel A MK-8266 0.7 /0.3 (Elderly Males With Mild/Mod. HTN) vs Panel A Placebo to MK-8266 (Elderly Males Mild/Moderate HTN); Test type: Other; p = 0.0019, ANOVA; Mean Difference (Final Values) = 7.79, 90% CI 2-sided [3.85 to 11.72]
Statistical Analysis 4: Comparison: Panel B MK-8266 0.3 mg (Elderly Females With Mild/Mod. HTN) vs Panel B Placebo to MK-8266 (Elderly Fem., Mild/Moderate HTN); Test type: Other; p = 0.2223, ANOVA; Mean Difference (Final Values) = 1.15, 90% CI 2-sided [-1.42 to 3.71]
Statistical Analysis 5: Comparison: Panel B MK-8266 0.6 mg (Elderly Females, Mild/Moderate HTN) vs Panel B Placebo to MK-8266 (Elderly Fem., Mild/Moderate HTN); Test type: Other; p = 0.0056, ANOVA; Mean Difference (Final Values) = 4.25, 90% CI 2-sided [1.69 to 6.82]
Statistical Analysis 6: Comparison: Panel B MK-8266 0.7/0.3 mg (Elderly Fem., Mild/Moderate HTN) vs Panel B Placebo to MK-8266 (Elderly Fem., Mild/Moderate HTN); Test type: Other; p = 0.0012, ANOVA; Mean Difference (Final Values) = 5.40, 90% CI 2-sided [2.83 to 7.96]

7. Primary Outcome: Number of Participants With Abnormal Electrocardiograms (ECG) Reported as an AE
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. An abnormal ECG value was any AE reported under the System Organ Classes of Investigations or Cardiac that was related to an abnormal ECG value.
Time Frame: Up to 48 days
Population: All participants who received at least one dose of the investigational drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Panel A MK-8266 0.3 mg (Elderly Males With Mild/Moderate HTN) | Panel A MK-8266 0.6 mg (Elderly Males With Mild/Moderate HTN) | Panel A MK-8266 0.7 /0.3 mg (Elderly Males, Mild/Moderate HTN) | Panel A Placebo to MK-8266 (Elderly Males, Mild/Moderate HTN) | Panel B MK-8266 0.3 mg (Elderly Females, Mild/Moderate HTN) | Panel B MK-8266 0.6 mg (Elderly Females, Mild/Moderate HTN) | Panel B MK-8266 0.7/0.3 mg (Elderly Fem., Mild/Moderate HTN) | Panel B Placebo to MK-8266 (Elderly Fem., Mild/Moderate HTN)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: MK-8266 Pharmacokinetic (PK) Parameter Area Under the Plasma Concentration Versus Time Curve From Time 0 Extrapolated to Infinity (AUC[0-inf])
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. (AUC[0-inf]) is a measure of the mean concentration levels of drug in the plasma after the dose.
Time Frame: Period 1, 2 and 3: Predose, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours postdose.
Population: The subset of participants who comply with the protocol sufficiently to ensure that these data will be likely to exhibit the effects of treatment, according to the underlying scientific model. AUC[0-inf] was not estimated for participants receiving placebo and for MK-8266 doses below 0.6 mg due to the lack of measureable concentrations.
Measure: Mean (Standard Deviation); unit: nM•hr
Arm/Group | Panel A MK-8266 0.3 mg (Elderly Males With Mild/Moderate HTN) | Panel A MK-8266 0.6 mg (Elderly Males With Mild/Moderate HTN) | Panel A MK-8266 0.7 /0.3 mg (Elderly Males, Mild/Moderate HTN) | Panel A Placebo to MK-8266 (Elderly Males, Mild/Moderate HTN) | Panel B MK-8266 0.3 mg (Elderly Females, Mild/Moderate HTN) | Panel B MK-8266 0.6 mg (Elderly Females, Mild/Moderate HTN) | Panel B MK-8266 0.7/0.3 mg (Elderly Fem., Mild/Moderate HTN) | Panel B Placebo to MK-8266 (Elderly Fem., Mild/Moderate HTN)
Number analyzed (Participants) | 0 | 6 | 6 | 0 | 0 | 6 | 6 | 0
nM•hr |  | 208 (81.5) | 314 (108) |  |  | 247 (66.8) | 449 (130) |
Statistical Analysis 1: Comparison: Panel A MK-8266 0.6 mg (Elderly Males With Mild/Moderate HTN) vs Panel B MK-8266 0.6 mg (Elderly Females, Mild/Moderate HTN); Test type: Other; GMR (Elderly female/Elderly male) = 1.23, 90% CI 2-sided [0.85 to 1.76] — GMR = geometric mean ratio

9. Secondary Outcome: MK-8266 PK Parameter Observed Maximum (Peak) Plasma Concentration (Cmax)
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. Cmax is a measure of the maximum amount of drug in the plasma after the dose is given.
Time Frame: Period 1, 2 and 3: Predose, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours postdose.
Population: The subset of participants who comply with the protocol sufficiently to ensure that these data will be likely to exhibit the effects of treatment, according to the underlying scientific model. Cmax was not estimated for participants receiving placebo.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Panel A MK-8266 0.3 mg (Elderly Males With Mild/Moderate HTN) | Panel A MK-8266 0.6 mg (Elderly Males With Mild/Moderate HTN) | Panel A MK-8266 0.7 /0.3 mg (Elderly Males, Mild/Moderate HTN) | Panel A Placebo to MK-8266 (Elderly Males, Mild/Moderate HTN) | Panel B MK-8266 0.3 mg (Elderly Females, Mild/Moderate HTN) | Panel B MK-8266 0.6 mg (Elderly Females, Mild/Moderate HTN) | Panel B MK-8266 0.7/0.3 mg (Elderly Fem., Mild/Moderate HTN) | Panel B Placebo to MK-8266 (Elderly Fem., Mild/Moderate HTN)
Number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 6 | 6 | 0
ng/mL | 7.76 (2.25) | 14.1 (3.45) | 16.2 (4.13) |  | 7.84 (1.80) | 17.8 (2.52) | 19.5 (2.61) |
Statistical Analysis 1: Comparison: Panel A MK-8266 0.3 mg (Elderly Males With Mild/Moderate HTN) vs Panel B MK-8266 0.3 mg (Elderly Females, Mild/Moderate HTN); Test type: Other; GMR (Elderly female/Elderly male) = 1.08, 90% CI 2-sided [0.88 to 1.33]
Statistical Analysis 2: Comparison: Panel A MK-8266 0.6 mg (Elderly Males With Mild/Moderate HTN) vs Panel B MK-8266 0.6 mg (Elderly Females, Mild/Moderate HTN); Test type: Other; GMR (Elderly female/Elderly male) = 1.26, 90% CI 2-sided [1.02 to 1.55]
Statistical Analysis 3: Comparison: Panel A MK-8266 0.7 /0.3 mg (Elderly Males, Mild/Moderate HTN) vs Panel B MK-8266 0.7/0.3 mg (Elderly Fem., Mild/Moderate HTN); Test type: Other; GMR (Elderly female/Elderly male) = 1.20, 90% CI 2-sided [0.98 to 1.48]

10. Secondary Outcome: MK-8266 PK Parameter Observed Time to Reach Cmax (Tmax)
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. Tmax is a measure of the time to reach the maximum concentration in the plasma after the drug dose. Nominal instead of actual times are presented.
Time Frame: Period 1, 2 and 3: Predose, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours postdose.
Population: The subset of participants who comply with the protocol sufficiently to ensure that these data will be likely to exhibit the effects of treatment, according to the underlying scientific model. Tmax was not estimated for participants receiving placebo.
Measure: Median (Full Range); unit: Hours
Arm/Group | Panel A MK-8266 0.3 mg (Elderly Males With Mild/Moderate HTN) | Panel A MK-8266 0.6 mg (Elderly Males With Mild/Moderate HTN) | Panel A MK-8266 0.7 /0.3 mg (Elderly Males, Mild/Moderate HTN) | Panel A Placebo to MK-8266 (Elderly Males, Mild/Moderate HTN) | Panel B MK-8266 0.3 mg (Elderly Females, Mild/Moderate HTN) | Panel B MK-8266 0.6 mg (Elderly Females, Mild/Moderate HTN) | Panel B MK-8266 0.7/0.3 mg (Elderly Fem., Mild/Moderate HTN) | Panel B Placebo to MK-8266 (Elderly Fem., Mild/Moderate HTN)
Number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 6 | 6 | 0
Hours | 2.0 [1.5 to 4.0] | 2.0 [1.5 to 3.0] | 2.0 [2.0 to 3.0] |  | 4.0 [2.0 to 6.0] | 3.5 [2.0 to 4.0] | 4.0 [3.0 to 12] |

11. Secondary Outcome: MK-8266 PK Parameter Apparent Half-Life (t1/2)
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. t1/2 is the time required for a given drug concentration in the plasma to decrease by 50%. Results are presented for the Harmonic Mean ± Pseudo standard deviation.
Time Frame: Period 1, 2 and 3: Predose, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours postdose.
Population: The subset of participants who comply with the protocol sufficiently to ensure that these data will be likely to exhibit the effects of treatment, according to the underlying scientific model. t1/2 was not estimated for participants receiving placebo and for MK-8266 doses below 0.6 mg due to the lack of measureable concentrations.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Panel A MK-8266 0.3 mg (Elderly Males With Mild/Moderate HTN) | Panel A MK-8266 0.6 mg (Elderly Males With Mild/Moderate HTN) | Panel A MK-8266 0.7 /0.3 mg (Elderly Males, Mild/Moderate HTN) | Panel A Placebo to MK-8266 (Elderly Males, Mild/Moderate HTN) | Panel B MK-8266 0.3 mg (Elderly Females, Mild/Moderate HTN) | Panel B MK-8266 0.6 mg (Elderly Females, Mild/Moderate HTN) | Panel B MK-8266 0.7/0.3 mg (Elderly Fem., Mild/Moderate HTN) | Panel B Placebo to MK-8266 (Elderly Fem., Mild/Moderate HTN)
Number analyzed (Participants) | 0 | 6 | 6 | 0 | 0 | 6 | 6 | 0
Hours |  | 12.7 (4.8) | 14.3 (3.8) |  |  | 13.6 (4.5) | 15.4 (3.4) |

12. Secondary Outcome: The Time Weighted Average Systolic Blood Pressure (SBP) Evaluated Over 8 Hours Post Dose (TWA[0-8hrs]) Following a Single Oral Dose of MK-8266.
Description: Participants rested for at least 10 minutes prior to having vital sign measurements obtained. Single dose effects on central SBP were estimated as a time-weighted average over the 8-hour post single dose observation period.
Time Frame: Up to 8 hours post dose in each dosing period (Up to 8 hours)
Population: The analysis population was all participants who received at least 1 dose of the investigational drug.
Measure: Least Squares Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Panel A MK-8266 0.3 mg (Elderly Males With Mild/Moderate HTN) | Panel A MK-8266 0.6 mg (Elderly Males With Mild/Moderate HTN) | Panel A MK-8266 0.7 /0.3 mg (Elderly Males, Mild/Moderate HTN) | Panel A Placebo to MK-8266 (Elderly Males, Mild/Moderate HTN) | Panel B MK-8266 0.3 mg (Elderly Females, Mild/Moderate HTN) | Panel B MK-8266 0.6 mg (Elderly Females, Mild/Moderate HTN) | Panel B MK-8266 0.7/0.3 mg (Elderly Fem., Mild/Moderate HTN) | Panel B Placebo to MK-8266 (Elderly Fem., Mild/Moderate HTN)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
millimeters of mercury | 146.4 (11.73) | 134.2 (12.96) | 132.7 (12.34) | 136.8 (8.61) | 142.4 (13.19) | 135.0 (8.22) | 136.0 (6.82) | 146.6 (12.54)
Statistical Analysis 1: Comparison: Panel A MK-8266 0.3 mg (Elderly Males With Mild/Moderate HTN) vs Panel A Placebo to MK-8266 (Elderly Males, Mild/Moderate HTN); Test type: Superiority; p = 0.0253, ANOVA; MK-8266 0.3 mg vs. placebo = 9.58, 90% CI 2-sided [1.69 to 17.46]
Statistical Analysis 2: Comparison: Panel A MK-8266 0.6 mg (Elderly Males With Mild/Moderate HTN) vs Panel A Placebo to MK-8266 (Elderly Males, Mild/Moderate HTN); Test type: Superiority; p = 0.2856, ANOVA; MK-8266 0.6 mg vs. placebo = -2.59, 90% CI 2-sided [-10.5 to 5.29]
Statistical Analysis 3: Comparison: Panel A MK-8266 0.7 /0.3 mg (Elderly Males, Mild/Moderate HTN) vs Panel A Placebo to MK-8266 (Elderly Males, Mild/Moderate HTN); Test type: Superiority; p = 0.1895, ANOVA; MK-8266 0.7 mg/ 0.3 mg vs. placebo = -4.06, 90% CI 2-sided [-11.9 to 3.82]
Statistical Analysis 4: Comparison: Panel B MK-8266 0.3 mg (Elderly Females, Mild/Moderate HTN) vs Panel B Placebo to MK-8266 (Elderly Fem., Mild/Moderate HTN); Test type: Superiority; p = 0.1157, ANOVA; MK-8266 0.3 mg vs. placebo = -4.16, 90% CI 2-sided [-10.0 to 1.70]
Statistical Analysis 5: Comparison: Panel B MK-8266 0.6 mg (Elderly Females, Mild/Moderate HTN) vs Panel B Placebo to MK-8266 (Elderly Fem., Mild/Moderate HTN); Test type: Superiority; p = 0.0018, ANOVA; MK-8266 0.6 mg vs. placebo = -11.7, 90% CI 2-sided [-17.5 to -5.79]
Statistical Analysis 6: Comparison: Panel B MK-8266 0.7/0.3 mg (Elderly Fem., Mild/Moderate HTN) vs Panel B Placebo to MK-8266 (Elderly Fem., Mild/Moderate HTN); Test type: Superiority; p = 0.0034, ANOVA; MK-8266 0.7 mg/ 0.3 mg vs. placebo = -10.6, 90% CI 2-sided [-16.5 to -4.77]

ADVERSE EVENTS:
Time Frame: Up to 48 days
Description: An adverse event (AE) is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
  The analysis population included all participants who received at least one dose of the investigational drug.
Arm/Group | Panel A MK-8266 0.3 mg (Elderly Males With Mild/Moderate HTN) | Panel A MK-8266 0.6 mg (Elderly Males With Mild/Moderate HTN) | Panel A MK-8266 0.7 /0.3 mg (Elderly Males, Mild/Moderate HTN) | Panel A Placebo to MK-8266 (Elderly Males, Mild/Moderate HTN) | Panel B MK-8266 0.3 mg (Elderly Females, Mild/Moderate HTN) | Panel B MK-8266 0.6 mg (Elderly Females, Mild/Moderate HTN) | Panel B MK-8266 0.7/0.3 mg (Elderly Fem., Mild/Moderate HTN) | Panel B Placebo to MK-8266 (Elderly Fem., Mild/Moderate HTN)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/6 | 4/6 | 3/6 | 1/6 | 5/6 | 4/6 | 4/6 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panel A MK-8266 0.3 mg (Elderly Males With Mild/Moderate HTN) (N=6) | Panel A MK-8266 0.6 mg (Elderly Males With Mild/Moderate HTN) (N=6) | Panel A MK-8266 0.7 /0.3 mg (Elderly Males, Mild/Moderate HTN) (N=6) | Panel A Placebo to MK-8266 (Elderly Males, Mild/Moderate HTN) (N=6) | Panel B MK-8266 0.3 mg (Elderly Females, Mild/Moderate HTN) (N=6) | Panel B MK-8266 0.6 mg (Elderly Females, Mild/Moderate HTN) (N=6) | Panel B MK-8266 0.7/0.3 mg (Elderly Fem., Mild/Moderate HTN) (N=6) | Panel B Placebo to MK-8266 (Elderly Fem., Mild/Moderate HTN) (N=6)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 2 (5)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.